CLINICAL TRIAL: NCT04023461
Title: Isolation of Pulmonary Veins With PVAC GOLD in Elderly Patients
Acronym: PVAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Mauricio Ibrahim Scanavacca, Arrhythmia Clinical Unit Director, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4471/16/137
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Atrial Fibrillation Paroxysmal; Cardiac Arrythmias
Keywords: Radiofrequency Ablation; Atrial Fibrilation; PVAC GOLD catheter; Elderly patients
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: All patients in clinical treatment arm had to keep on antiarrhythmic drug for AF rhythm control strategy
Who Masked: Care Provider, Outcomes Assessor
Masking Description: At the time of patient recruitment, they were randomly assigned to ablation or medical therapy (antiarrhythmic drug arm) according to a 1:1 stratified randomization list locked into a computer system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Treatment Group (No Intervention)
- Interventional Ablation Group (Experimental)
  Interventions: Device: PVAC GOLD catheter ablation

INTERVENTIONS:
Device: PVAC GOLD catheter ablation — Isolation of pulmonary veins using PVAC GOLD catheter.
  Arms: Interventional Ablation Group

SUMMARY:
It is a prospective, randomized and double-blind clinical trial involving an invasive technique for isolation of pulmonary veins (PVAC gold) in relation to clinical treatment during an one year of segment. The patients included have paroxysmal atrial fibrillation (aged 65 years and older) refractory to antiarrhythmic treatments that do not have structural and / or ischemic heart diseases. This trial employed quality of life scores prior to the study and during the sixth and twelfth month of the segment, electrocardiograms and holter of 24 hours. The proposed imaging tests was the transesophageal echocardiogram before each procedure. The cerebral MRI was performed in the 24 hours post invasive procedure and Angio-tomography of the pulmonary veins in the 6-month segment.

DETAILED DESCRIPTION:
Objective: Pulmonary vein isolation (PVI) for atrial fibrillation (AF) has become progressively safer and more effective with advances in single-shot devices. The aim of this study was to compare catheter ablation (CA) of second-generation pulmonary vein ablation catheter (PVAC) Gold technique versus clinical treatment in elderly patients (≥ 65 years old) with symptomatic paroxysmal AF (PAF) without structural heart diseases.

Methods: Prospective randomized study that selected consecutive patients with paroxysmal atrial fibrillation older than 65 years-old in two groups: (1) PVAC ablation group and (2) antiarrhythmic drugs therapy group. Primary outcomes were AF recurrences, progression to persistent AF forms. As secondary outcomes, changes in Mini-Mental State Examination and AF Quality of Life Score were accessed.This study doesn't include payment of participants. All patients signed the informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Indication for isolation of pulmonary veins
* Age >= 65 years old
* Association with the following characteristics:

  1. Symptomatic Atrial Fibrillation;
  2. Sinusal Rhythm maintenance failure for at least 1 Antiarrythmic Drugs;
  3. Diagnosis of Atrial Fibrilation on resting eletrocardiogram and/or 24h Holter.

Exclusion Criteria:

* Prior Atrial Fibrillation ablation;
* Atrial Fibrillation permanent and/or persistent;
* Left atrial size > 55 mm;
* Mechanical prothetic mitral valve replacement;
* Presence of atrial thrombus;
* Cardiac invasive procedure < 90 days;
* Cerebral embolism < 6 months;
* Hypertrophic cardiomyopathy;
* Contraindications to antiocoagulation and cerebral MRI.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Recurrence of atrial fibrillation | 1 year after ablation
  Recurrence of atrial fibrillation during 1 year of follow-up

SECONDARY OUTCOMES:
Occurrence of Asymptomatic Cerebral Embolism | 1 year of follow-up
  Occurrence of Asymptomatic Cerebral Embolism during 1 year of follow-up
Esophageal Ulcer | 24 hours after pulmonary vein isolation
  Esophageal Ulcer documented by Esophagus-gastro-duodenoscopy after ablation procedure
Quality of Life Assessment | 1 year after ablation
  Quality of Life in Atrial Fibrillation Questionnaire Score

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio I Scanavacca, MD, PhD, Principal Investigator — Arrythmia Clinical Unit Director
Locations (1):
- Arrhythmia Clinical Unit - Instituto do Coração - HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No